CLINICAL TRIAL: NCT00912743
Title: A Phase II, Open-Label, Multicenter Trial to Assess the Efficacy and Safety of the PARP Inhibitor, Olaparib, Alone in Previously-Treated Patients With Stage IV, Measurable Colorectal Cancer, Stratified by MSI Status
Brief Title: Efficacy and Safety of Olaparib in Pretreated Patients With Measurable Colorectal Cancer, Stratified by Microsatellite Instability (MSI) Status
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9010C00008; AGICC 09CRC01
Record Dates: First submitted 2009-05-28; First posted 2009-06-03 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Olaparib; MSI status; Stage IV; Measurable Colorectal Cancer; Stratified by MSI Status
MeSH Terms: conditions — Colorectal Neoplasms | interventions — olaparib

ARMS (1):
- 1 (Experimental): MSI - H arm
  Interventions: Drug: olaparib

INTERVENTIONS:
Drug: olaparib — 400 mg po bid continuously

SUMMARY:
This study is being carried out to see if the new drug, olaparib (AZD2281), can effectively and safely treat advanced large bowel cancer. The primary goal of this clinical trial is to determine whether olaparib will have a beneficial effect on the patient's cancer by causing a response and increasing the time it takes for the cancer to progress.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have measurable disseminated colorectal cancer that is incurable by surgery
* Patients will have had tumor progression following standard combination front-line or second-line chemotherapy.
* CRC patients who have relapsed or recurrent disease within six months after completing adjuvant or neoadjuvant chemotherapy

Exclusion Criteria:

* Previous treatment with PARP inhibitors, including olaparib.
* Patients with symptomatic, uncontrolled brain metastases.
* Patients receiving any chemotherapy, radiotherapy (except for palliative reasons), within 4 weeks from the last dose prior to study entry (or a longer period depending on the defined characteristics of the agents used).
* Patients who are unable to swallow orally administered medication.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence P Leichman, MD, Principal Investigator — Aptium Oncology Gastrointestinal Cancer Consortium; Bert H O'Neil, MD, Principal Investigator — Aptium Oncology Gastrointestinal Cancer Consortium; Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca
Locations (8):
- United States (8):
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, Aurora, Colorado
  - Research Site, Newark, Delaware
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Seattle, Washington

REFERENCES:
- See also: CSR_Synopsis_D9010C00008 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=638&filename=D9010C00008.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Target accrual: 54 subjects. MSI-H group: 15; non-MSI-H group: 39. Pre-planned interim analysis of the non-MSI-H cohort, after 17 patients, stopped recruitment into that cohort. Recruitment to the MSI-H cohort continued.
Pre-assignment Details: Subjects with stage IV, measurable disseminated CRC incurable by surgery, with tumour progression following standard combination front-line or second-line chemotherapy, relapsed or recurrent disease within 6 months completing adjuvant or neoadjuvant chemotherapy and met all inclusion/exlusion criteria.
Groups:
- MSI-H: MSI-H group receiving olaparib 400mg BID
- Non-MSI-H: Non-MSI-H group receiving olaparib 400mg BID
Period: Overall Study
Arm/Group | MSI-H | Non-MSI-H
Started | 13 | 20
Completed | 0 | 0
Not Completed | 13 | 20
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 9 | 18
Not completed — Toxicity | 0 | 1
Not completed — End of treatment form was not collected | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSI-H | Non-MSI-H | Total
Number analyzed (Participants) | 13 | 20 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) at screening
  years | 51.77 (9.37) | 61.80 (11.46) | 57.85 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender, Male/Female
  Participants
    Female | 6 | 9 | 15
    Male | 7 | 11 | 18
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    White | 10 | 19 | 29
    Black or African American | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Tumour Response
Description: Tumour response is the number of patients who experienced complete or partial response at least once during the assessment period, according to the definitions of Response Evaluation Criteria In Solid Tumours (RECIST version 1.1)
Time Frame: From baseline, i.e. up to 28 days before first study drug dose, and then every 2 cycles (8 weeks) up to objective disease progression by RECIST, assessed up to 35 months
Population: Full analysis set - all treated patients
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MSI-H | Non-MSI-H
Number analyzed (Participants) | 13 | 20
Percentage of Participants | 0 [0 to 25] | 0 [0 to 17]

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the duration from first dose till objective progression or death. In absence of progression or death, the time is calculated from first dose till last evaluable scanning visit.
Time Frame: as for outcome 1
Population: Full analysis set - all treated patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MSI-H | Non-MSI-H
Number analyzed (Participants) | 13 | 20
days | 61 [52 to 360] | 55 [49 to 56]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration from first dose till death from any cause. In absence of death, the time is calculated from first dose till the date subject last known to be alive
Time Frame: Survival follow-up from first dose till death of the patient or till end of study in absence of death, assessed up to 35 months
Population: Full analysis set - all treated patients
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MSI-H | Non-MSI-H
Number analyzed (Participants) | 13 | 20
days | 248 [121 to 554] | 290.5 [157 to 429]

ADVERSE EVENTS:
Arm/Group | MSI-H | Non-MSI-H
Serious Adverse Events (participants affected / at risk) | 6/13 | 3/20
Other Adverse Events (participants affected / at risk) | 12/13 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSI-H (N=13) | Non-MSI-H (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vena cava injury (Injury, poisoning and procedural complications) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MSI-H (N=13) | Non-MSI-H (N=20)
Anaemia (Blood and lymphatic system disorders) | 6 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 8 | 15
Vomiting (Gastrointestinal disorders) | 6 | 9
Fatigue (General disorders) | 5 | 8
Oedema peripheral (General disorders) | 2 | 4
Blood creatinine increased (Investigations) | 2 | 2
Haemoglobin decreased (Investigations) | 1 | 3
Anorexia (Metabolism and nutrition disorders) | 3 | 5
Dizziness (Nervous system disorders) | 3 | 1
Dysgeusia (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2
Chills (General disorders) | 1 | 2
Oedema (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 3 | 0
Nocturia (Renal and urinary disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less